CLINICAL TRIAL: NCT04913298
Title: Prospective Quality Assurance Study for the Application of Cytosorb® in Patients With Cytokine Storm, Rhabdomyolysis and Acute Liver Failure
Brief Title: Prospective Study for the Application of Cytosorb® in Critically Ill Patients
Acronym: Cyto-SOLVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Michael Zoller MD, Principle Investigator, Ludwig-Maximilians - University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-0236
Record Dates: First submitted 2021-05-07; First posted 2021-06-04 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Rhabdomyolysis; Acute Liver Injury; Cytokine Storm
Keywords: Cytosorb; adsorption kinetics; saturation; critically ill patients
MeSH Terms: conditions — Rhabdomyolysis; Cytokine Release Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cytosorb therapy (Other): blood samples are taken before and after the cytokine adsorber at given times
  Interventions: Device: Cytosorb therapy

INTERVENTIONS:
Device: Cytosorb therapy — Start of Cytosorb therapy is at the discretion of the attending physician

SUMMARY:
The mortality of critically ill patients is persistently high and requires targeted therapy of pathophysiological disorders. One approach to optimize therapy is the use of the cytokine adsorber Cytosorb®, which has a CE certification for the indications hyperinflammation, rhabdomyolysis and liver failure and is therefore frequently used in patients with sepsis, polytrauma and acute liver failure. Although few clinical data describe the efficiency mostly retrospectively, there are no data on real-time elimination performance and saturation kinetics during the course of treatment. These questions should be answered by the present study.

ELIGIBILITY:
Inclusion Criteria:

* intensive care therapy
* hyperinflammation or acute liver dysfunction or rhabdomyolysis
* need of continuous renal replacement therapy
* treatment with Cytosorb (decision of the attending physician)

Exclusion Criteria:

- other reasons for Cytosorb application

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Change (percentage) in different cytokines (measured as a cytokine panel) measured pre- and post-CytoSorb® (extracorporeal) in intensive care patients with hyperinflammation | 12 hours
  Measurement of a cytokine panel (20 different cytokines in one panel) before and after the filter at different times.
Change (percentage) in myoglobin measured pre- and post-CytoSorb® (extracorporeal) in intensive care patients with rhabdomyolysis | 12 hours
  Measurement of myoglobin before and after the filter at different times.
Change (percentage) in bile acids (measured as a panel) measured pre- and post-CytoSorb® (extracorporeal) in intensive care patients with acute liver failure | 12 hours
  Measurement of bile acids before and after the filter at different times.

SECONDARY OUTCOMES:
Change (percentage) in norepinephrine demand before and after the use of CytoSorb® | 2 years
Change ( percentage ) of liver toxic substances (e.g. bile acids) in patients´ blood due to the use of CytoSorb® | 2 years
Change ( percentage ) of myoglobin in patients´ blood due to the use of CytoSorb® | 2 years
Difference (percentage) between predicted mortality and real mortality of patients treated with CytoSorb® | 2 years
  Mortality can be predicted by intensive care scores. We will investigate the difference between actual and predicted mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- LMU munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Graf H, Grafe C, Bruegel M, Happich FL, Wustrow V, Wegener A, Wilfert W, Zoller M, Liebchen U, Paal M, Scharf C. Extracorporeal Elimination of Pro- and Anti-inflammatory Modulators by the Cytokine Adsorber CytoSorb(R) in Patients with Hyperinflammation: A Prospective Study. Infect Dis Ther. 2024 Sep;13(9):2089-2101. doi: 10.1007/s40121-024-01028-8. Epub 2024 Aug 18. PMID 39154299
- [Derived] Graf H, Grafe C, Bruegel M, Zoller M, Maciuga N, Frank S, Weidhase L, Paal M, Scharf C. Myoglobin adsorption and saturation kinetics of the cytokine adsorber Cytosorb(R) in patients with severe rhabdomyolysis: a prospective trial. Ann Intensive Care. 2024 Jun 22;14(1):96. doi: 10.1186/s13613-024-01334-x. PMID 38907120
- [Derived] Greimel A, Habler K, Grafe C, Maciuga N, Brozat CI, Vogeser M, Zoller M, Happich FL, Liebchen U, Frank S, Paal M, Scharf C. Extracorporeal adsorption of protective and toxic bile acids and bilirubin in patients with cholestatic liver dysfunction: a prospective study. Ann Intensive Care. 2023 Nov 9;13(1):110. doi: 10.1186/s13613-023-01198-7. PMID 37943350